CLINICAL TRIAL: NCT00220220
Title: Efficacy and Safety of Amlodipine Used as add-on Therapy in Moderately to Severely Hypertensive Patients Not Adequately Controlled by Olmesartan Medoxomil 20 mg Monotherapy
Brief Title: Amlodipine as add-on to Olmesartan in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS8663-A-E302
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2007-10

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Amlodipine

INTERVENTIONS:
Drug: olmesartan medoxomil
Drug: amlodipine

SUMMARY:
Test the efficacy and safety of the combination of olmesartan and amlodipine in hypertensive patients whose blood pressure is not adequately controlled with olmesartan alone.

ELIGIBILITY:
Inclusion Criteria:

* Mean sitting BP of greater than or equal to 140/90-115 mmHg and mean 24h dBP greater than or equal to 80 mmHg with at least 30% of daytime readings greater than 85 mmHg prior to randomization.

Exclusion Criteria:

* Secondary hypertension of any aetiology;
* Any serious disorders which may limit the ability to evaluate the efficacy or safety of the test drug(s);
* History of myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, congestive heart failure, hypertensive encephalopathy, stroke or TIA within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Mean change in trough sitting diastolic blood pressure (dBP) assessed by conventional BP measurements after 8 weeks of double-blind treatment.

SECONDARY OUTCOMES:
Mean change in trough sitting sBP and mean BP daytime, nighttime and 24h ABPM after 8 weeks of double-blind treatment.
Responder rate, defined as number (%) of patients achieving BP goals during 8 weeks of double-blind treatment.
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brommer, MD, Principal Investigator
Locations (6):
- Germany (6):
  - Hamburg
  - Magdeburg
  - Messkirch
  - Stuhr
  - Tann
  - Worpswede

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Barrios V, Brommer P, Haag U, Calderon A, Escobar C. Olmesartan medoxomil plus amlodipine increases efficacy in patients with moderate-to-severe hypertension after monotherapy: a randomized, double-blind, parallel-group, multicentre study. Clin Drug Investig. 2009;29(7):427-439. doi: 10.2165/00044011-200929070-00001. PMID 19499960